CLINICAL TRIAL: NCT06691230
Title: PeRfusiOn Post tHrombEcTomy (PROPHET) A Prospective Observational Cohort Study
Brief Title: PeRfusiOn Post tHrombEcTomy (PROPHET)
Acronym: PROPHET
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-01108
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Stroke, Acute, Ischemic
Keywords: Acute ischemic stroke; Large-vessel occlusion; Endovascular mechanical thrombectomy; Flat-panel detector computed tomography perfusion imaging; Perfusion imaging
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Flat-panel detector computed tomography perfusion imaging, FDCTP: Potential clinical use of FDCTP acquired during or shortly after the endovascular stroke treatment

SUMMARY:
Endovascular mechanical thrombectomy is the standard of care for treating patients with a large-vessel occlusion acute ischemic stroke. However, in more than half of these patients, remaining distal vessel occlusions limit the benefit of this therapy. Currently the detection of residual vessel occlusions and the decision for further treatment by the operator is based on the 2D digital subtraction angiography (DSA) images. However, this technique has several limitations. Recently, a new imaging technique, with the possibility to acquire 3D time-resolved perfusion images directly in the operating room was introduced (the flat-panel detector computed tomography perfusion imaging, FDCTP). It can overcome the spatial limitations of 2D DSA, but the details on clinical validation and utility of FDCTP are currently lacking.

DETAILED DESCRIPTION:
This clinical investigation is planned as a multi-center, prospective, non-randomized observational study with a primary endpoint to evaluate a potential diagnostic benefit. The diagnostic tool to be studied is clinically indicated 60s Dyna CT Head Perfusion (FDCTP imaging) obtained after or during mechanical thrombectomy for acute ischemic stroke.

The population consists of patients with symptoms of acute ischemic stroke, who were intended to undergo mechanical thrombectomy. This means that patients who did not undergo mechanical thrombectomy and only had diagnostic angiography (e.g. physician team has decided against thrombectomy due to pre-interventional vessel reperfusion), can still be included in the study. Patients can only be included if a FDCTP was acquired immediately after thrombectomy or diagnostic angiography by the treating physician team as part of the standard clinical routine. There is no control group.

The overall objective is to investigate the potential clinical use of FDCTP acquired during or shortly after the endovascular stroke treatment. Primary study objective is to evaluate in how many cases FDCTP maps reveal new, potentially relevant clinical information that may change treatment decisions. The primary research hypothesis is that the proportion of patients where FDCTP reveals new, potentially clinically relevant findings is greater than 25%. Assuming a true proportion of 33% of the primary outcome, we will need 251 patients to reach a power of 80% at a one-sided alpha of 2.5%, based on a one-sample binomial exact test. To account for a drop-out rate of 10%, we plan to recruit 279 patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by a signature
* The patients received mechanical thrombectomy or there was the intention to perform endovascular treatment, but only diagnostic angiography was performed.
* Patients received FDCTP as clinically indicated by the treating physician.

Exclusion Criteria:

* Inability to give consent due to insufficient knowledge of the project language
* Inability to follow the clinically indicated visit at 90 days after the index stroke (e.g. patients living abroad).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an acute ischemic stroke with large vessel occlusion who have undergone endovascular mechanical thrombectomy and received a (flat-panel detector computed tomography perfusion imaging (FDCTP) shortly after the treatment.
Sampling Method: Probability Sample
Enrollment: 279 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Detection of New Potentially Clinically Relevant Findings on FDCTP | Up to 30 days post-procedure
  * Any hypoperfusion on processed FDCTP maps suggesting residual vessel occlusion within the target mechanical thrombectomy territory, not noted on the 2D DSA imaging (dichotomous variable: yes versus no)
  * Any hypoperfusion suggestive of vessel occlusion outside the target mechanical thrombectomy territory not observed on the 2D DSA i.e., a new vessel occlusion (dichotomous variable: yes versus no)
  * No hypoperfusion suggestive of residual vessel occlusion on FDCTP within the target mechanical thrombectomy territory, even thought the patient has incomplete reperfusion (<eTICI3) on the 2D DSA (dichotomous variable: yes versus no)
  The primary outcome of the study will be assessed as a dichotomous variable (yes versus no), derived from a compound measure of clinically relevant findings based on the three interpretations described above.

SECONDARY OUTCOMES:
Diagnostic Sensitivity of 2D DSA vs. FDCTP in Detecting Residual Vessel Occlusion | Up to 30 days post-procedure
  Proportion of patients with all detected residual vessel occlusions on FDCTP versus none or not all detected residual vessel occlusions on FDCTP (dichotomous outcome)

OTHER OUTCOMES:
Eloquence of Hypoperfused Tissue | Up to 30 days post-procedure
  Hypoperfusion in the eloquent brain zones i.e. eloquent cortex (dichotomous variable: yes versus no)
Concordance between FDCTP and standard imaging | Up to 30 days post-procedure
  Association of findings from the FDCTP with standard cross-sectional imaging on follow-up examination at 24 hours (categorical variable: sustained reperfusion, persisting perfusion deficit, delayed reperfusion)
Prevalence of the No-Reflow Phenomenon on FDCTP | Up to 30 days post-procedure
  Proportion of patients with/without residual microvascular hypoperfusion (dichotomous variable).
Detection of Competitive Leptomeningeal Flow on FDCTP | Up to 30 days post-procedure
  American Society of Interventional and Therapeutic Neuroradiology Collateral Grading System (categorical variable, Score 0-4)
Cost-effectiveness of FDCTP | Up to 30 days post-procedure
  Incremental cost-effectiveness ratio (ICER, continuous variable)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Kaesmacher, Prof., Principal Investigator — University of Bern
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Basel
  - University Hospital Bern, Bern

IPD SHARING:
Plan to Share IPD: Undecided